CLINICAL TRIAL: NCT03864263
Title: The Prevalence of Hepatitis B Virus Infection in Immunized Children With HBsAg-positive Parents
Brief Title: Hepatitis B Virus Infection in Immunized Children With HBsAg-positive Parents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qiu Li (Other)
Responsible Party: Sponsor-Investigator, Qiu Li, Children's Hospital of Chongqing Medical University, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Other Study IDs: 2019-30
Record Dates: First submitted 2019-03-04; First posted 2019-03-06 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Hepatitis b Virus Infection
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with HBsAg-positive patients: Children from a father or mother who are infected with HBV
- Children without a family history of HBV: Children without a family history of HBV infection

INTERVENTIONS:
Other:

SUMMARY:
Hepatitis B virus (HBV) infection is a major public health problem facing the world, with more than 2 billion people infected with HBV. There are more than 400 million chronic carriers, and 75% of carriers live in the Asia Pacific region.

The mother-to-child transmission route of hepatitis B virus is recognized as one of the most important routes of transmission, and recent studies have found that fathers who are carriers of HBV may also be one of the risk factors for HBV infection in children, but as far as the investigators know. Therefore, as a high-population area in China, the purpose of this study is to investigate the prevalence of HBV infection in this population.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) infection is a major public health problem facing the world, with more than 2 billion people infected with HBV. Although since 1986 the World Health Organization (WHO has reduced the incidence of hepatitis B virus-related chronic liver disease, cirrhosis and hepatocellular carcinoma by incorporating hepatitis B vaccination into routine vaccination programmes for infants and adolescents, There are more than 400 million chronic carriers, and 75% of carriers live in the Asia Pacific region. Occult hepatitis B virus infection (OBI) is HBV surface antigen negative, but HBV DNA can be detected by PCR. Although the clinical consequences of OBI have not yet been fully determined, recent studies have shown that OBI may cause HBV-related diseases such as hepatitis B, cirrhosis, hepatocellular carcinoma, or aggravation or aggravation, and patients who receive immunosuppression through organ or blood transfusion. OBI reactivation has occurred. The protective effect on humans after vaccination with hepatitis B vaccine has the investigator sakened over time, and anti-HBs-negative children may have a higher risk of HBV infection due to loss of protection.

The mother-to-child transmission route of hepatitis B virus is recognized as one of the most important routes of transmission, and recent studies have found that fathers who are carriers of HBV may also be one of the risk factors for HBV infection in children, but as far as the investigators know, only Studies in Taiwan and other places have reported studies on HBV infection in children with HBV-infected mothers, and no research has focused on the effects of fathers' HBV positivity on children. Therefore, as a high-population area in China, the purpose of this study is to investigate the prevalence of HBV infection in this population.

ELIGIBILITY:
Inclusion Criteria:

* The father or (and) mother is HBV-infected (pre-pregnancy or present)；
* Children is vaccinated with hepatitis B vaccine after birth;

Exclusion Criteria:

* Children with HBV infection;
* Participants agreed to undergo clinical follow-up studies.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The father or (and) mother is a HBV-infected person (pre-pregnancy or present), who is vaccinated with hepatitis B vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-07-04 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of hepatitis b virus infection | 0-5 years
  Clinical follow-up testing for "overt" or "occult" HBV infection in immunized Children With HBsAg-positive Parents

CONTACTS AND LOCATIONS:
Overall Officials: Yao Zhao, Principal Investigator — Chongqing Children's Hospital of Chongqing Medical University
Locations (1):
- Chongqing Children's Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: Undecided